CLINICAL TRIAL: NCT06221215
Title: Clinical Analysis of the Hormone Between Patients With Moderate and Severe Traumatic Brain Injury and Cerebral Hemorrhage
Brief Title: Clinical Analysis of Early Hormones Between Patients With Traumatic Brain Injury and Cerebral Hemorrhage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: GHNingxia
Record Dates: First submitted 2023-12-30; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Brain Injury Traumatic Diffuse With Loss of Consciousness
Keywords: Traumatic brain injury; Cerebral hemorrhage; hormone; trauma
MeSH Terms: conditions — Brain Injuries, Traumatic; Cerebral Hemorrhage; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Traumatic brain injury Group: The levels of related hormones (growth hormone, pituitary prolactin, ACTH, cortisol, FSH, thyroid hormone, etc.) were measured in patients with traumatic brain injury on the 1st, 7th and 14th day.
  Interventions: Procedure: trauma
- Spontaneous cerebral hemorrhage roup: The levels of related hormones (growth hormone, pituitary prolactin, ACTH, cortisol, FSH, thyroid hormone, etc.) were measured in patients with spontaneous craniocerebral injury on the 1st, 7th and 14th day.

INTERVENTIONS:
Procedure: trauma — The main purpose of this study is to observe whether the early hormone changes and trends in the two groups of patients with or without trauma.
  Groups: Traumatic brain injury Group

SUMMARY:
Our understanding of neurosecretory dysfunction after TBI is still insufficient, and the number of patients with neuroendocrine dysfunction caused by craniocerebral trauma may be underestimated, especially the neuroendocrine changes related to HPA axis in the early stage after craniocerebral trauma. Moreover, there are few and fragmentary literature data on the benefits of hormone replacement therapy in patients with neuroendocrine disorders after traumatic brain injury. This requires more studies to further determine the characteristics of pituitary function or hormone disorders in the early stage after traumatic brain injury, which makes it necessary for us to further study the neuroendocrine dysfunction (hormone disorder) in the early stage after craniocerebral injury. To explore the relationship between craniocerebral injury and early hormone disorder by measuring the changes of early hormone levels in patients with TBI is of great significance for the early detection of related complications after craniocerebral injury and the evaluation of the prognosis of patients with craniocerebral injury, and can provide a new diagnosis and treatment plan for early intervention of related complications after TBI.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. The patient was clearly diagnosed as craniocerebral injury.
3. The Glasgow score on admission was 3-12 (moderate and severe).
4. It has complete preclinical data.

Exclusion Criteria:

1. Complicated with other severe visceral injuries or severe systemic fractures.
2. Suffered from craniocerebral tumors, endocrine diseases, cardiovascular diseases, depression, sleep and mental disorders.
3. In the past month, there are people who receive immune and hormone therapy.
4. Women during pregnancy and lactation.
5. Where there is a logical or common sense error in the data entered.
6. The lack of too much clinical data related to this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Qualified inpatients hospitalized in our hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of GH | 1st, 7th and 14th day.
  The levels of related hormones (growth hormone) were measured in patients with TBI.
Change of pituitary prolactin | 1st, 7th and 14th day.
  The levels of related hormones (pituitary prolactin) were measured in patients with TBI.
Change of ACTH | 1st, 7th and 14th day.
  The levels of related hormones ( ACTH) were measured in patients with TBI.
Change of cortisol | 1st, 7th and 14th day.
  The levels of related hormones (cortisol) were measured in patients with TBI.
Change of FSH | 1st, 7th and 14th day.
  The levels of related hormones (FSH) were measured in patients with TBI.
Change of thyroid hormone | 1st, 7th and 14th day.
  The levels of related hormones (thyroid hormone) were measured in patients with TBI.

CONTACTS AND LOCATIONS:
Overall Officials: Zhanfeng Niu, Doctor, Study Director — General Hospital of Ningxia Medical University
Locations (1):
- The General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: Undecided